CLINICAL TRIAL: NCT04033692
Title: Post-market Clinical Follow-Up Study to Collect Safety, Performance and Clinical Benefits Data of the JuggerKnot Mini Soft Anchor for Use in the Maxillofacial Treatment of Temporomandibular Joint (TMJ)
Brief Title: MDR-JuggerKnot Mini Soft Anchor in Maxillofacial TMJ
Status: Withdrawn | Type: Observational
Why Stopped: Manufacturer decided not to proceed with study.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-64SM
Record Dates: First submitted 2019-07-18; First posted 2019-07-26 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: TMJ Disc Disorder; TMJ Pain; TMJ Sounds on Opening/Closing the Jaw; TMJ Disease
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- JuggerKnot Mini Soft Anchors: Patients who have been implanted with the JuggerKnot Mini Soft Anchor who have undergone repair, repositioning or reattachment of soft tissues, ligament and tendons to the mandible is require for surgical stabilization of the TMJ articular disc
  Interventions: Device: JuggerKnot Mini Soft Anchor

INTERVENTIONS:
Device: JuggerKnot Mini Soft Anchor — Patient who have been implanted with one or more JuggerKnot Mini Soft Anchor(s) who have undergone repair, repositioning or reattachment of soft tissues, ligament and tendons to the mandible is require for surgical stabilization of the TMJ articular disc.

SUMMARY:
The objective of this retrospective consecutive series PMCF study is to collect data confirming safety, performance and clinical benefits of the JuggerKnot Mini Soft Anchor (implant and instrumentation) when used for soft tissue to bone fixation in the treatment of temporomandibular joint (TMJ) surgery. Safety, performance, and clinical benefits will be evaluated at the following time points: pre op, 6 weeks, 3 months and 1-year follow-up. JuggerKnot Mini has been on the market since November of 2011.

DETAILED DESCRIPTION:
The primary objective is to confirm safety of the study products. This will be assessed by recording the incidence and frequency of revisions, complications, and adverse events. Relationship of the events to either implant or instrumentation should be specified.

The secondary objective is the assessment of performance and clinical benefits by analyzing recorded patient-reported clinical outcomes measures (PROMs).

ELIGIBILITY:
Inclusion Criteria:

* Implanted with one or more JuggerKnot Mini Soft Anchor(s) with either a 2-0 or 3-0 suture
* Must have undergone repair, repositioning or reattachment of soft tissues, ligament and tendons to the mandible is required for surgical stabilization of the TMJ articular disc

Exclusion Criteria:

* Local Infection.
* Patient conditions including blood supply limitations and insufficient quantity or quality off bone or soft tissue.
* Patients with mental or neurological conditions who are unwilling or incapable of following postoperative care instructions or patients who are otherwise unwilling or incapable of doing so.
* Foreign body sensitivity where material sensitivity is suspected.
* Off-label use.
* Sepsis.
* Patient is a prisoner.
* Patient is a known alcohol or drug abuser.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive series of subjects implanted with one or more JuggerKnot Mini Soft Anchors in the treatment of temporomandibular joint (TMJ) disease according to the approved indications for 93 total joints. Inclusion/exclusion criteria mirror the indications and contraindications in the IFU.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Device Safety Assessed Through the Incidence and Frequency of Revisions, Complications, and Adverse Events | Out to a minimum of 1 year
  Assessment of safety by recording and analyzing the incidence and frequency of revisions, complications, and adverse events.

SECONDARY OUTCOMES:
Device performance and Clinical Benefits Assessed by a Pain Assessment. and Temporomandibular Joint Function of the Pain Assessment Survey Case Report Form. | Out to a minimum of 1 year
  Pain Assessment is used to evaluate a patients pain from 0 to 10, 0 representing no pain at all and 10 representing the worse pain imaginable.
Device performance and Clinical Benefits Assessed by a TMJ Function Pain Assessment Survey Case Report Form | Out to a minimum of 1 year
  The TMJ Function portion of the Pain Assessment Survey is assessed by if the patient experiences Temporomandibular Joint Clicking or Popping Noise. The Joint Clicking or Popping noise is evaluated as a Yes the joint click when opening and closing the mouth, or No the joint does not click when opening and closing the mouth on either the left or right side.
Device performance and Clinical Benefits Assessed by a Headache Pain Assessment Survey Case Report Form | Out to a minimum of 1 year
  The Headache portion of the Pain Assessment Survey is evaluated as, Yes the patient has headaches, or No the patient does not have headaches. If they check yes the survey asks on which side of the headache occurs and in which location. Location options are: Front, Posterior, Temporal or Top of the head.

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, Study Director — Zimmer Biomet

IPD SHARING:
Plan to Share IPD: No